CLINICAL TRIAL: NCT05961033
Title: The Effects of Virtual Reality Based Exercises on Pain, Range of Motion and Quality of Life in Patients With Adhesive Capsulitis
Brief Title: The Effects of Virtual Reality Based Exercises in Patients With Adhesive Capsulitis
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Collaborators: Sakarya University of Applied Sciences (Unknown)
Responsible Party: Principal Investigator, Oguzhan Bahadir DEMIR, Principal Investigator, Kocaeli University
Other Study IDs: 32/22
Record Dates: First submitted 2023-06-26; First posted 2023-07-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2023-08

CONDITIONS: Pain; Quality of Life; Range of Motion; Virtual Reality
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study: Individuals in the first group to be included in the study group will be included in a virtual reality-based exercise program for half an hour a day, 5 days a week for a total of 4 weeks, in addition to routine electrotherapy programs for half an hour a day, 5 days a week for a total of 4 weeks. These individuals will be able to play the games saved in the Oculus Quest 2 SG system in the virtual environment, thanks to the three-dimensional glasses and handpiece that can be worn on the head.
  Interventions: Device: Virtual Reality based exercises
- control: Individuals who receive traditional electrotherapy and exercise program

INTERVENTIONS:
Device: Virtual Reality based exercises — Play VR games
  Groups: study

SUMMARY:
Musculoskeletal disorders such as adhesive capsulitis (AC) affect tissues such as muscles, bones, joints, tendons and ligaments and are the second most disabling condition worldwide. Musculoskeletal Systemic disorders are typically characterized by pain, limitations in joint range of motion or functional ability.

Existing studies have shown that Virtual Reality (VR) is beneficial in pain management for example; pain relief during dressing changes in burn patients. VR can also reduce anxiety, distract from the fear of pain, and reduce stress. It can distract the patients who are afraid of moving due to pain and enable them to move freely. In this study, AC patients will be treated with VR application. Patients pain levels, upper extremity range of motion, functional activity levels and quality of life levels will be evaluated. A total of 36 patients will be included in the study.

This observational randomized controlled study will contribute to the literature by investigating the effects of VR based exercises in individuals with AC.

DETAILED DESCRIPTION:
Individuals in the first group to be included in the study group will be included in a VR-based exercise program for half an hour a day, 5 days a week for a total of 4 weeks, in addition to routine electrotherapy programs for half an hour a day, 5 days a week for a total of 4 weeks. These individuals will use the Oculus Quest 2 VR system in the virtual environment thanks to the three-dimensional glasses and handpiece that can be worn on the head. They will play the registered games. These games will include purpose-oriented activities such as lying on the head and using bilaterally, which are intended to use the upper extremities of individuals with AC in daily life. Participants will be treated under the constant supervision of a physiotherapist, will be rested at the end of the exercise, and will leave the clinic after making sure that there is no problem.

Individuals in the second group, who will be included in the traditional exercise group, will be included in the stretching and strengthening exercise program for half an hour a day, 5 days a week for a total of 4 weeks, for a total of 10 hours, in addition to the routine electrotherapy programs for half an hour a day, 5 days a week for a total of 4 weeks. The exercises will be performed by a physiotherapist working in the clinic and blind to the study.

Pain levels (Visual Analogue Scale), upper extremity range of motion (Goniometric measurement), functional activity levels (Shoulder Pain and Disability Index) and quality of life (SF-36) of all participants will be evaluated before and after the study.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Clinical diagnosis of adhesive capsulitis

Exclusion Criteria:

* Inability to cooperate VR
* Surgery on the upper extremity or trunk
* Neurological disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed as having Adhesive Capsulitis and being treated in the rehabilitation center
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Pain severity change | Initial assessment before playing VR exercises, secondary assessment after 4 weeks VR based exercises
  pain intensity after VR based exercises will be assessed by Visual Analogue Scale (VAS). VAS is often used to measure the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain (0-10). Ten shows more pain intensity.
Quality of Life level change | Initial assessment before playing VR exercises, secondary assessment after 4 weeks VR based exercises
  Level of Quality of Life will be assessed by Short Form- 36 (SF-36). SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and have been widely used. High points show high quality ol life levels.
Shoulder functionality level change | Initial assessment before playing VR exercises, secondary assessment after 4 weeks VR based exercises
  Shoulder functionality will be assessed by Shoulder and Pain Disability Inventory (SPADI). The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder. The means of the two subscales are averaged to produce a total score ranging from 0 (best) to 100 (worst).

SECONDARY OUTCOMES:
Shoulder mobility angles change | Initial assessment before playing VR exercises, secondary assessment after 4 weeks VR based exercises
  Shouder mobility will be assessed by goniometric measurement

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Kocaeli University Faculty of Medicine Hospital, Kocaeli
  - Sakarya University Physiotherapy and Rehabilitation Research Center, Sakarya

IPD SHARING:
Plan to Share IPD: No